CLINICAL TRIAL: NCT01560468
Title: Phase I Study of Hepatitis C Virus (HCV) Entry Inhibitor (ITX 5061) in Liver Transplant Recipients With HCV Infection
Brief Title: Study of Hepatitis C Virus (HCV) Entry Inhibitor in Liver Transplant Recipients With HCV Infection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Financial Reasons
Sponsor: Schiano, Thomas D., MD (Other)
Collaborators: iTherX Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSM 12-00045; 12-0123 (Other: Mount Sinai GCO)
Record Dates: First submitted 2012-02-15; First posted 2012-03-22 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Hepatitis C Infection
Keywords: Hepatitis C Virus Infection; Liver Transplantation
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ITX 5061 (Experimental): Subjects will receive ITX 5061 for 28 days beginning at the time of liver transplantation for hepatitis C virus. 300mg will be administered on the day of surgery and for one week post transplant, followed by 150mg for an additional 21 days.
  Interventions: Drug: ITX 5061

INTERVENTIONS:
Drug: ITX 5061 — 300 mg given orally beginning at the time of liver transplantation and for 1 week post-transplant followed by 150 mg orally for an additional 21 days.

SUMMARY:
This study will test the safety and tolerability of HCV Entry Inhibitor ITX 5061 in Liver Transplant Recipients with Hepatitis C infection. The investigators hypothesize that ITX 5061 oral monotherapy will be safe in adults during and after liver transplantation and that therapy will also inhibit HCV infection of newly transplanted livers in adults with prior HCV infection.

DETAILED DESCRIPTION:
All subjects will receive 28 days of ITX 5061 beginning at the time of transplant.

Dosing of ITX 5061 is as follows:

Day of Transplant prior to surgery: ITX 5061 300 mg Day of Transplant following surgery: ITX 5061 300 mg Post-Operative Days 1-6: ITX 5061 300 mg Post-Operative Days 7-27: ITX 5061 150 mg

Subjects will be monitored for HCV RNA levels, HDL cholesterol and ITX 5061 drug concentration levels.

A liver biopsy will be performed at 6 months post-transplant to assess for histological signs of HCV recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-72
* Patients accepted onto waiting list for liver transplantation for HCV related liver disease and receiving a deceased donor liver allograft
* HCV RNA (+) at time of listing for transplantation. All HCV genotypes will be eligible
* Patients with HCC and those receiving hepatitis B core (+) donor livers will be eligible
* Standard immunosuppression protocol with tacrolimus, corticosteroid taper, and mycophenolate mofetil

Exclusion Criteria:

* Viral co-infection (HBV/HIV)
* Receipt of a HCV (+) donor allograft
* Patients undergoing retransplantation for recurrent HCV
* Multivisceral transplantation
* Patients receiving anti-viral therapy at the time of LT
* Live donor liver transplantation

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-03; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Incidence of HCV recurrence post-transplant | 28 days
  We hypothesize that ITX 5061 oral monotherapy will be safe in adults during and after liver transplantation and will inhibit HCV infection of newly transplanted livers in adults with prior HCV infection. The number of treated subjects who are infected at 28 days post-transplant will be compared to the historical control rate (95%).

SECONDARY OUTCOMES:
Change in serum HCV RNA | 3 months after transplant
  To determine the change in serum HCV RNA from study entry to end of dosing (28 days) and 3 month follow up
Levels of ITX 5061 | 28 days
  To assess trough levels of plasma ITX 5061 throughout the dosing period
Viral dynamics of serum HCV RNA | 24 hours post-transplant
  To characterize the viral dynamics of serum HCV RNA levels during the first 24 hours post-transplant
Potential changes in plasma HCV E2 | 28 days
  To characterize potential changes in plasma HCV E2 (HCV envelope protein) regions in the setting of ITX 5061 administration

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Schiano, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Sulkowski MS, Kang M, Matining R, Wyles D, Johnson VA, Morse GD, Amorosa V, Bhattacharya D, Coughlin K, Wong-Staal F, Glesby MJ; AIDS Clinical Trials Group A5277 Protocol Team. Safety and antiviral activity of the HCV entry inhibitor ITX5061 in treatment-naive HCV-infected adults: a randomized, double-blind, phase 1b study. J Infect Dis. 2014 Mar 1;209(5):658-67. doi: 10.1093/infdis/jit503. Epub 2013 Sep 16. PMID 24041792